CLINICAL TRIAL: NCT04717297
Title: A Tailored Medication Management Intervention for Older Adults
Brief Title: Tailored Medication Management Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Emily Somerville, Instructor of Occupational Therapy and Neurology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202008139
Record Dates: First submitted 2021-01-13; First posted 2021-01-22 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Medication Non Adherence; Polypharmacy
Keywords: Medication Management; Occupational Therapy; Older adults
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tailored Medication Management Remote Intervention Treatment Arm (Experimental): Participants receive a total of three visits (one evaluation/pre-treatment visit and 2 treatment visits) that last 75 minutes each over 4 weeks. Sessions/visits are spaced 1 week apart and will be delivered remotely.
  Interventions: Behavioral: Medication Management Remote Intervention
- Waitlist Attention Control Arm (Sham Comparator): The attention control group will receive two, 75-minute attention visits with a trained research assistant. Upon completion of waitlist period, the participants in the waitlist group will be offered the intervention in person.
  Interventions: Behavioral: Waitlist Control
- Tailored Medication Management In-Person Intervention Treatment Arm (Experimental): Participants receive a total of three visits (one evaluation/pre-treatment visit and 2 treatment visits) that last 75 minutes each over 4 weeks. Sessions/visits are spaced 1 week apart and will be delivered in-person.
  Interventions: Behavioral: Medication Management In-Person Intervention

INTERVENTIONS:
Behavioral: Medication Management Remote Intervention — First, the study pharmacist reviews the older adult's medication for potentially inappropriate medications. The pharmacist collaborates with the prescribing physician(s) to deprescribe as indicated. The pharmacist educates the older adult and OT on any changes that were made. The OT and older adult will develop a plan to reduce risk factors and improve medication management. Participants receive tailored compensatory strategies and supports to remediate extrinsic risk factors and modify the home environment to improve medication adherence. The OT provides training and active practice of the compensatory strategies and supports in the home in an effective and safe manner. All components of the intervention will be delivered remotely.
  Arms: Tailored Medication Management Remote Intervention Treatment Arm
Behavioral: Waitlist Control — A trained research assistant will complete two attention control visits in the homes of participants. Visit will consist of semi-structured interview exploring the participant's life history.
  Arms: Waitlist Attention Control Arm
Behavioral: Medication Management In-Person Intervention — Participants in the waitlist control will be offered the medication management intervention to be completed in person. If they consent, the study pharmacist will review their medication for potentially inappropriate medications. The pharmacist will collaborate with the prescribing physician(s) to deprescribe any inappropriate medication as indicated. The pharmacist will educate the older adult and OT on any changes. The OT and older adult will develop a plan to reduce risk factors and improve medication management. Participants will receive tailored compensatory strategies and supports to remediate extrinsic risk factors and modify the home environment to improve medication adherence. The OT will provide training and active practice of the compensatory strategies and supports in the home in an effective and safe manner. All components of the intervention will be delivered in person.
  Arms: Tailored Medication Management In-Person Intervention Treatment Arm

SUMMARY:
Successful medication management is an essential instrumental activity of daily living (IADL) for older adults with polypharmacy; however, between 40%-70% of older adults fail to take their medications as prescribed. Providing interventions to address medication management and restore performance for this IADL is within the scope of practice for occupational therapy (OT), however, there is paucity of evidence for OT interventions to improve medication management in community-dwelling older adults. We have developed a tailored medication management intervention (TIMM) for community-dwelling older adults which recognizes the unique context in which medication management occurs (the home) and addresses the personal and environmental barriers experienced by older adults. TIMM is delivered in the home, by an OT, and in collaboration with a pharmacist to reduce inappropriate polypharmacy.

DETAILED DESCRIPTION:
Almost 70% of older adults experience multimorbidity and medication is often the first intervention used to manage it. In fact, 90% of older adults take at least one medication and 36% take 5 or more, commonly known as polypharmacy. When taken correctly, medication can extend life-expectancy and improve quality of life. However, estimates show 40-75% of community-dwelling older adults are nonadherent, or deviate from their medication regimen. These older adults are at an increased risk of nonadherence because the physical changes associated with multimorbidity including decreased memory, fine motor skills, and visual acuity and because of the complexity polypharmacy adds to a medication routine. Nearly 43% of older adults with polypharmacy take medications that are inappropriate and can cause negative long term physical and cognitive function, which further complicates the mediation management process.

Nonadherence has significant consequences which include increased health care costs, falls, institutionalization, and decreased medication effectiveness, quality of life. In fact, improving medication adherence has been identified as a public health concern by the World Health Organization. Despite this, interventions designed to improve adherence in older adults remain largely ineffective. The majority of interventions are disease or medication specific or are implemented with a "one size fits all" approach (e.g. providing standard pill organizers that may be difficult for some older adults to open). Furthermore, interventions are often implemented in a clinical setting such as doctor's office or hospital and do not consider the unique home environment where medication management typically occurs. Home environments can offer support (i.e. caregiver to set up medications) or barriers (i.e. low lighting that makes medications difficult to see) to medication management. Given the complexity of each older adult's risk factors and home environment, a more tailored, individualized approach must be considered.

Tailored, individualized interventions aimed at remediating the environmental barriers in the home have been successful in improving daily activity performance for older adults. However, this type of intervention has not been tested specifically to improve medication adherence in older adults with multimorbidity and polypharmacy. We propose a tailored, individualized medication management intervention (TIMM) for community-dwelling older adults with multimorbidity and polypharmacy. TIMM is an interdisciplinary, compensatory intervention which consists of: 1) an initial in-home evaluation of medication management ability, individual risk factors, and identification of environmental barriers to independence; 2) a medication review by a pharmacist to address polypharmacy; and 3) tailored intervention by an occupational therapist to improve adherence by reducing barriers to medication management.

We will conduct an equivalency randomized control trial to examine the feasibility, acceptability and preliminary efficacy of TIMM delivered remotely and in-person. The use of telehealth to deliver occupational therapy interventions for older adults has become more widely utilized, especially during the last two years. Remote interventions remove many of the barriers to in-home care including access and cost and have been shown to be an effective delivery method for OT and other medical services for older adults. Participants in the treatment group will receive the intervention delivered remotely, and participants in the waitlist control group will receive the intervention in-person, upon completion of their control period.

ELIGIBILITY:
Inclusion Criteria:

* 65 and older
* takes 5 or more medications
* Decreased medication adherence (one or more "yes" responses on Medication Adherence Rating Scale (MARS))

Exclusion Criteria:

* Cognitive impairment as indicated by Short Blessed Test (SBT) score of 10 or more
* Lives in institutional setting

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Recruitment | 6 months
  Recruitment and retention rate
Dose | 6 months
  Treatment minutes and number of treatment sessions
Treatment Fidelity | 6 months
  Ability to deliver required treatment session elements
Intervention Safety- ER Visits | 6 months
  Number of ER visits
Intervention Safety- Hospitalizations | 6 months
  Number of unplanned hospitalizations
Intervention Safety- Doctor Visits | 6 months
  Number of unplanned doctor visits
Intervention Safety- Falls | 6 months
  Number of falls
Intervention Safety | 6 months
  Number of therapy visits
Intervention Pharmacy Cost | 6 months
  Pharmacist time
Intervention OT Cost | 6 months
  OT time
Intervention Modification Cost | 6 months
  adaptive equipment cost

SECONDARY OUTCOMES:
Medication Management Ability | 6 months
  In-Home Medication Management Evaluation (HOME-Rx) which includes measures of ability to independently manage mediations and barriers to medication management
Potentially Inappropriate Medications | 6 months
  BEERS Criteria for Inappropriate Medication Use in Older Patients
Equivalency | 6 months
  Equivalency of remote vs in person intervention on all primary outcome measures

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Somerville E, Bollinger R, Keleman A, Haxton M, Sarrami B, Chen SW, Holden B, Yan Y, Stark S. Tailored medication management intervention delivered by occupational therapists for older adults: A study protocol. Br J Occup Ther. 2023 Apr;86(4):257-264. doi: 10.1177/03080226221135366. Epub 2023 Mar 21. PMID 40337485

DOCUMENTS (1):
  • Informed Consent Form (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT04717297/ICF_000.pdf